CLINICAL TRIAL: NCT04207658
Title: The Effects Of Pushing Techniques During Second Stage Of Labour
Brief Title: The Effects Of Pushing Techniques During Second Stage Of Labour On Maternal and Newborn Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Evrim Bayraktar, Assoc Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ERU
Record Dates: First submitted 2019-11-08; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Prevention; Newborn Complication
Keywords: pushing technıques; maternal health; fetal health

STUDY DESIGN:
Intervention Model Description: The data of the study is collected by using Baseline Obstetric Data Form in which demographic, obstetric, and first stage features of labour with features of 2nd, 3rd and 4th stages of pregnancy are registered, and Visual Analogue Fatigue Scale (VAFS).
  .Management of Data Collection Tools and Forms Randomization of gravitas participated in the study is done with the help of computers. The second stage of labour is defined as the time passed after the cervical dilatation reaches 10cm. The expulsion stage is the time between the sight of baby's head in the vulva and the end of labour.
  The pushing is initiated; when the servical dilatation is 10cm along with strong uterus contractions until foetal head rotation is over and when the foetal head is at least "+1" in the pelvis. In addition, at the onset of pushing in spontaneous group, woman's desire to push is not ignored.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valsalva's Pushing (Experimental): The gravitas are informed about spontaneous pushing at the active phase of dilatation (6cm) in second stage of labour and they are encouraged for spontaneous pushing just at the onset of pushing. At the expulsion phase (baby's head is visible in vulva), they are encouraged to perform the Valsalva's manoeuvre that they have practised in routines of delivery; When contractions start, breathe twice normally. Take a deep breath and hold. Compress the air with the help of diaphragm and abdominal muscles. Push strongly and long (for 10-15 sec). Breathe out and take another deep breath, hold it and push as strongly as possible for another 10-15 seconds. Stop pushing when contractions are mild. Breathe 2-3 times in normal style. Relax and have a rest until the next contraction.
  Interventions: Behavioral: Valsalva's Style Pushing
- control (No Intervention): Practices on Spontaneous Pushing Group The gravitas are informed about spontaneous pushing at the active phase of dilatation (6cm) in second stage of labour and they are encouraged for spontaneous pushing just at the onset of pushing. Just after feeling the push, the gravitas are requested perform pushing as follows; Breathe normally until participants feel the push when contractions start, pull back muscles surrounding the uterus while breathing. Start pushing gradually and breathe out smoothly by minimizing lips. Push between breaths for 5-6 seconds while pushing downwards by breathing out. Breathe normally when contractions weaken.

INTERVENTIONS:
Behavioral: Valsalva's Style Pushing — The second stage of labour is defined as the time passed after the cervical dilatation reaches 10cm. The expulsion stage is the time between the sight of baby's head in the vulva and the end of labour. the participants are given information about the study after self introduction of each gravid is done for completing baseline obstetric data forms by midwives. Also, blood samples for pre and postpartum haemoglobin level changes are collected. The perineal area is examined for postpartum tears through pad checks. Vital findings (respiration, pulse and TA) are evaluated prior to their transfer to the delivery room. Just after the birth, mothers are tested for pH, pO2, pCO2 and lactate levels in blood while the newborns are tested for pH, pO2 (mmHg) and pCO2 levels through umbilical artery along with 1st min and 5 min APGAR analysis. The visual scale is utilized for determination of first 24-hour fatigue and they are recorded in follow-up forms.
  Arms: Valsalva's Pushing

SUMMARY:
Purpose :To determine the impact of directed Valsalva's's versus spontaneous pushing techniques during second stage of labour on postpartum maternal fatigue. .

Methods: The control group participants have an onset of spontaneous pushing when the cervical dilatation was 6cm while the directed pushing group carried out the Valsalva's manoeuvre.The data of the study are obtained by utilizing Baseline Obstetric Data Form and Visual Analogue Fatigue Scale (VAFS). The investigators have done postpartum tests on perineal tear, hemorrhagia, haemoglobin level, vital findings, blood pH, pO2 and pCO2, and lactate level for the mother while the neonatal tests of APGAR score for 1st and 5th minutes, umbilical artery blood pH, pO2 and pCO2 levels are done for the newborn.

DETAILED DESCRIPTION:
Vaginal births are often associated with some form of trauma to the genital tract, and tears that affect the anal sphincter or mucosa (third- and fourth-degree tears) can cause serious problems. Perineal trauma can occur spontaneously or result from a surgical incision (episiotomy). Different perineal techniques are being used to slow down the birth of the baby's head, and allow the perineum to stretch slowly to prevent injury. Massage, warm compresses and different perineal management techniques are widely used by midwives and birth attendants.

A computer program designed by an independent group of the clinical research centre is creating the randomisation list, in blocks of four to six (randomly chosen by the electronic system and well balanced by centre) and stratified by maternity ward and within maternity wards by both parity (nulliparous vs multiparous) and epidural analgesia use at randomisation. The randomisation and the data collection will be performed at a website available 24 hours a day.

After the midwives-investigators have verified the inclusion and exclusion criteria and collected the signed informed consent, the randomisation will take place. There is no conceivable way to conduct this study on either a double-blinded or single-blinded basis.

Sample The population of our study consists of primigravida hospitalized at Erciyes University Training and Research Hospital. In line with data in the literature, the computations are done considering the fulfilment rate of Valsalva's Manoeuvre pushing as 20% and 50% in spontaneous pushing for fewer interventions through wellness of baby and the mother. Thus, sample volumes to represent the population are p1= 0.20 (control group), p2= 0.50 (experimental group), %95 confidence interval, α= 0.05, β = 0.20, power = 0.80 (1-β) for each group n=82 women, and in total 164 mothers.

Criteria of primigravida in the study; Women are accepted in the study on condition that they are aged 18 and more, primigravida, bearing single foetus between 2500 and 3999gr of birth weight in vertex position, in 38-42 gestation weeks, expected to have spontaneous vaginal labour with no or little risk factors, without obstetrical or medical complications during labour, with a cervical dilatation of 6cm and an amnion sack opening at 3cm of cervical dilatation, and they must also accept to participate in the study.

Practices on Spontaneous Pushing Group The gravitas are informed about spontaneous pushing at the active phase of dilatation (6cm) in second stage of labour and they are encouraged for spontaneous pushing just at the onset of pushing. Just after feeling the push, the gravitas are requested perform pushing as follows; Breathe normally until participants feel the push when contractions start, pull back muscles surrounding the uterus while breathing. Start pushing gradually and breathe out smoothly by minimizing lips. Push between breaths for 5-6 seconds while pushing downwards by breathing out. Breathe normally when contractions weaken.

Practices on Valsalva's Style Pushing Group The gravitas are informed about spontaneous pushing at the active phase of dilatation (6cm) in second stage of labour and they are encouraged for spontaneous pushing just at the onset of pushing. At the expulsion phase (baby's head is visible in vulva), they are encouraged to perform the Valsalva's manoeuvre that they have practised in routines of delivery; When contractions start, breathe twice normally. Take a deep breath and hold. Compress the air with the help of diaphragm and abdominal muscles. Push strongly and long (for 10-15 sec). Breathe out and take another deep breath, hold it and push as strongly as possible for another 10-15 seconds. Stop pushing when contractions are mild. Breathe 2-3 times in normal style. Relax and have a rest until the next contraction.

Data collection tools and forms The data of the study is collected by using Baseline Obstetric Data Form in which demographic, obstetric, and first stage features of labour with features of 2nd, 3rd and 4th stages of pregnancy are registered, and Visual Analogue Fatigue Scale (VAFS).

.Management of Data Collection Tools and Forms Randomization of gravitas participated in the study is done with the help of computers. The second stage of labour is defined as the time passed after the cervical dilatation reaches 10cm. The expulsion stage is the time between the sight of baby's head in the vulva and the end of labour.

The pushing is initiated; when the servical dilatation is 10cm along with strong uterus contractions until foetal head rotation is over and when the foetal head is at least "+1" in the pelvis. In addition, at the onset of pushing in spontaneous group, woman's desire to push is not ignored.

The practices on gravids of our study (spontaneous and Valsalva's pushing) are applied as follows;

• The participants are given information about the study after self introduction of each gravid is done for completing baseline obstetric data forms by midwives. Also, blood samples for pre and postpartum haemoglobin level changes are collected. The perineal area is examined for postpartum tears through pad checks. Vital findings (respiration, pulse and TA) are evaluated prior to their transfer to the delivery room. Just after the birth, mothers are tested for pH, pO2, pCO2 and lactate levels in blood while the newborns are tested for pH, pO2 (mmHg) and pCO2 levels through umbilical artery along with 1st min and 5 min APGAR analysis. The visual scale is utilized for determination of first 24-hour fatigue and they are recorded in follow-up forms.

Data Assessment The obtained data is assessed through SPSS 22.0 (Statistical Package of Social Science). While assessing these data, along with descriptive statistical methods, tests that are appropriate for data distribution in comparison of quantitative data (mean, standard deviation or median) are utilized. The results are assessed in 95% confidence interval and p<0.05 meaningful.

2.7 Data Analysis Shapiro-Wilk's test was used, histograms and q-q plots were also assessed to test the data normality. Levene test was used to assess variance homogeneity. For comparisons, either two-sided independent samples t test or Mann-Whitney U test was used for continuous variables and chi-square analysis were used for categorical variables. Values are expressed n(%), mean±SD or median(25th-75th percentiles). All analysis were performed using R 3.2.1 (www.r-project.org) software. A p value less than 5% was considered as statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Women are accepted in the study on condition that they are aged 18 and more
* Primigravida
* bearing single foetus between 2500 and 3999gr of birth weight in vertex position
* in 38-42 gestation weeks
* they must also accept to participate in the study
* with a cervical dilatation of 6cm

Exclusion Criteria:

* obstetrical or medical complications during labour,
* expected to have spontaneous vaginal labour with risk factors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
Women with valsalva pushing in upright position during second stage of labor will have proper fetal wellbeing than those with spontaneous pushing stage of labor duration and maternal and fetal arterial blood gas tests. | 15 minutes from birth
  Just after the birth, mothers are tested for pH, pO2, pCO2 and lactate levels in blood while the newborns are tested for pH, pO2 (mmHg) and pCO2 levels through umbilical artery
Women with valsalva pushing in upright position during second stage of labor will have proper fetal wellbeing than those with spontaneous pushing stage of labor duration and maternal postpartum hemorrhage | 24 hours from birth.
  The perineal area is examined for postpartum tears through pad checks.
Women with valsalva pushing in upright position during second stage of labor will have proper fetal wellbeing than those with spontaneous pushing stage of labor duration and newborn APGAR scores. | 1st min and 5 minutes from birth.
  1st min and 5 min APGAR analysis for newborn
Women with valsalva pushing in upright position during second stage of labor will have proper fetal wellbeing than those with spontaneous pushing stage of labor duration and maternal vital finding. | 24 hours from birth.
  Vital findings (respiration, pulse and TA) are evaluated prior to their transfer to the delivery room.
Women with valsalva pushing in upright position during second stage of labor will have proper fetal wellbeing than those with spontaneous pushing stage of labor duration and maternal haemoglobin level. | 6 and 24 hours from birth.
  Blood samples for pre and postpartum haemoglobin level changes are collected.

SECONDARY OUTCOMES:
Women with spontaneous pushing in upright position during second stage of labor will have proper fetal wellbeing than those with valsalva pushing stage of labor duration and maternal haemoglobin level. | 6 and 24 hours from birth.
  Blood samples for pre and postpartum haemoglobin level changes are collected.
Women with spontaneous pushing in upright position during second stage of labor will have proper fetal wellbeing than those with valsalva pushing stage of labor duration and maternal and fetal arterial blood gas tests. | 15 minutes from birth
  just after the birth, mothers are tested for pH, pO2, pCO2 and lactate levels in blood while the newborns are tested for pH, pO2 (mmHg) and pCO2 levels through umbilical artery
Women with spontaneous pushing in upright position during second stage of labor will have proper fetal wellbeing than those with valsalva pushing stage of labor duration and maternal postpartum hemorrhage | 24 hours from birth.
  The perineal area is examined for postpartum tears through pad checks.
Women with spontaneous pushing in upright position during second stage of labor will have proper fetal wellbeing than those with valsalva pushing stage of labor duration and newborn APGAR analysis | 1st min and 5 minutes from birth.
  1st min and 5 min APGAR analysis for newborn
Women with spontaneous pushing in upright position during second stage of labor will have proper fetal wellbeing than those with valsalva pushing stage of labor duration and maternal Vital findings. | 24 hours from birth.
  Vital findings (respiration, pulse and TA) are evaluated prior to their transfer to the delivery

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Bayraktar, Principal Investigator — Erciyes Üniversitesi Sağlık Bilimleri Fakültesi
Locations (1):
- Evrim Bayraktar, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided